CLINICAL TRIAL: NCT00100321
Title: Immunologic Studies of Tumors of the Pancreas
Brief Title: Surgery for Pancreatic Tumors and Collection of Tumor Tissue for Study
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050044; 05-C-0044; NCT00104832 (obsolete NCT alias)
Record Dates: First submitted 2004-12-28; First posted 2004-12-29 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-11-20

CONDITIONS: Pancreatic Neoplasms
Keywords: Tumor Antigen Identification; Standard Treatment; Tissue Acquisition; Surgery; Adjuvant Chemotherapy; Pancreatic Cancer; Pancreatic Tumor
MeSH Terms: conditions — Pancreatic Neoplasms

SUMMARY:
This study will examine pancreatic tumor tissue and immune cells from patients with a pancreatic tumor to look for markers on these cells that may be useful in developing new treatments for the disease.

Patients 16 years of age and older with any evidence of a primary pancreatic tumor that can be surgically removed may be eligible for this study. Types of pancreatic tumors included in this trial are pancreatic cancer, adenosquamous carcinoma, anaplastic carcinoma, IPMN (intraductal pancreatic mucinous neoplasm), acinar cell carcinoma, pancreaticoblastoma, mucinous cystic neoplasms, serous cystic neoplasms, solid-pseudopapillary cystic neoplasms, squamous cell carcinoma, Vater (ampullary tumors) duodenal adenoma or cancer and common bile duct tumors (cholangiocarcinoma.) The specific type of tumor does not have to be determined before the operation. Candidates are screened with a medical history and physical examination, computed tomography (CT) or magnetic resonance imaging (MRI) of the chest, abdomen, and pelvis, blood and urine tests, and an electrocardiogram. Patients older than 50 years of age and patients with a history of cardiovascular disease may also have a thallium cardiac stress test.

Participants undergo standard treatment for their pancreatic tumor, including surgery to remove the tumor. Before, during, and after the operation, several blood samples are drawn as part of routine patient care and for research tests. During the surgery, a small piece of tumor tissue is taken for examination under the microscope and to grow cells in the laboratory for tumor and immune cell studies. Some patients may undergo leukapheresis to collect large numbers of white blood cells for study. For this procedure, blood is collected through a needle in an arm vein and flows through a catheter (plastic tube) into a machine that separates it into its components by centrifugation (spinning). The white cells are extracted and the rest of the blood (plasma, red cells, and platelets) is returned through another needle in the other arm.

Patients who require additional treatment, such as chemotherapy or radiation, may be treated at NIH on another protocol or referred for appropriate treatment elsewhere.

DETAILED DESCRIPTION:
Background:

* Effective standard treatment options are currently not available for exocrine pancreas carcinomas. Adenocarcinoma of the pancreas, the most frequent exocrine tumor, is the fourth leading cause of cancer related deaths in men or women in this country.
* Immunotherapy for melanoma as studied in the Surgery Branch has resulted in striking tumor regression in some patients.
* Procurement of lymphocytes and tumor from patients with pancreas cancer will facilitate the identification of tumor-associated antigens leading to rational extensions of adoptive therapy and vaccination directed against this disease.

Objectives:

* Primary Objective: To obtain tissue, both tumor and lymphocytes, which can be used to identify tumor antigens specific to the various histologies of pancreas and ampullary cancer along with the HLA restricted epitopes of these antigens.
* Secondary Objective: To treat patients with resectable pancreas neoplasms using standard pancreatic resection and follow for survival.

Eligibility:

* Any patient greater than or equal to16 years of age with radiographic or endoscopic evidence of a pancreatic mass, ampullary mass or malignant stricture without evidence of distant metastases
* Patients must have an ECOG performance score of 0-2.
* Patients must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to biopsy or surgery.

Design:

* A tissue acquisition trial in which tissues will be obtained at the time of surgical operation for the resection of pancreas exocrine tumors.
* Tissue will be processed by the Surgery Branch Cell processing lab in accordance with their standard practices.
* No investigational therapy will be given.
* It is anticipated that 180 patients will be enrolled over 7 years.

ELIGIBILITY:
* INCLUSION CRITERIA

Any patient greater than or equal to 16 years of age with radiographic or endoscopic evidence of a pancreatic mass, ampullary mass or malignant stricture without evidence of distant metastases.

Recovered from any serious toxicity experienced during previous treatment (chemo-, radiation, hormone, immuno-, etc., therapy) for pancreas cancer to a grade 2 or less.

ECOG Performance Status greater 0-2.

Must have laboratory and physical examination parameters within acceptable limits by standard of practice guidelines prior to surgery.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-12-21; Study Completion 2012-11-20

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Murray T, Samuels A, Ghafoor A, Ward E, Thun MJ. Cancer statistics, 2003. CA Cancer J Clin. 2003 Jan-Feb;53(1):5-26. doi: 10.3322/canjclin.53.1.5. PMID 12568441
- [Background] Parkin DM, Bray FI, Devesa SS. Cancer burden in the year 2000. The global picture. Eur J Cancer. 2001 Oct;37 Suppl 8:S4-66. doi: 10.1016/s0959-8049(01)00267-2. No abstract available. PMID 11602373
- [Background] Abbruzzese JL. New applications of gemcitabine and future directions in the management of pancreatic cancer. Cancer. 2002 Aug 15;95(4 Suppl):941-5. doi: 10.1002/cncr.10753. PMID 12209675